CLINICAL TRIAL: NCT03542955
Title: The Efficacy/Safety Profile Of Pulsed Shortwave Therapy in Cervical Osteoarthritis: A Comparison Study Against Etoricoxib
Brief Title: Pulse Shortwave Therapy in Cervical Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioElectronics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO180402
Record Dates: First submitted 2018-05-16; First posted 2018-06-01 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2018-05

CONDITIONS: Cervical Osteoarthritis
MeSH Terms: interventions — Etoricoxib; Analgesics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ActiPatch Group (Active Comparator): Subjects in this group will receive an active pulsed shortwave therapy device to wear 24 hours a day for 4 weeks.
  Interventions: Device: ActiPatch
- Control Group (Placebo Comparator): Subjects in this group will take Etoricoxib 60mg, once daily for 4 weeks.
  Interventions: Drug: Etoricoxib 60 mg

INTERVENTIONS:
Device: ActiPatch — A Pulsed Shortwave Therapy Device
  Other Names: pulsed shortwave therapy
  Arms: ActiPatch Group
Drug: Etoricoxib 60 mg — nonsteroidal anti-inflammatory drug used as standard therapy
  Other Names: analgesic
  Arms: Control Group

SUMMARY:
The ActiPatch is an FDA cleared pain therapy device that uses pulsed shortwaves to interrupt pain signals at the nerve. 200 patients will be randomized and divided into an ActiPatch treatment group and comparison analgesic drug therapy group . Subjects will be assessed with the Neck Disability Index (NDI) at baseline and at four weeks and VAS scores will be recorded in order to determine the efficacy of the ActiPatch device compared to Etoricoxib. Cervical osteoarthritis causes chronic neck pain which could potentially be alleviated by the ActiPatch without the use of medication.

DETAILED DESCRIPTION:
Cervical Osteoarthritis causes chronic pain in the neck due to the discs of the spine breaking down, losing fluid, and becoming stiffer over time. As obesity and age increase, the likelihood of cervical osteoarthritis increases as well. When the pain caused by the broken down discs becomes severe, it may result in a loss of mobility in the neck region. Chronic neck pain has a serious impact on not only quality of life, but can also negatively affect a persons ability to lead a healthy active lifestyle. Standard analgesic therapy it limited in efficacy and can result in serious adverse effects specially with long term use.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Neck Pain of > 2 months
* Cervical Osteoarthritis - Radiological Evidence
* Males & females
* Age: 30-60 years

Exclusion Criteria:

* Neck Pain <2 months
* Pregnancy
* Irreversible neck injury
* Congenital Neurological/Muscular Diseases
* Osteo-articular Disorders
* Auto-immune Diseases
* Osteoporosis
* Hematological Diseases (Thalassemia/Sickle Cell Anemia)
* Cancer
* Contra-indication to Etoricoxib 60 mg
* Age <30 or >60 years

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | 4 weeks
  It is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. The NDI has sufficient support and usefulness to retain its current status as the most commonly used self-report measure for neck pain.
  The NDI can be scored as a raw score or doubled and expressed as a percent. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. Al the points can be summed to a total score. The test can be interpretated as a raw score, with a maximum score of 50, or as a percentage. A higher score indicates more patient-rated disability.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 4 weeks
  Visual analog scale [VAS] is a measure of pain intensity. It is a continuous scale comprised of a horizontal (called horizontal visual analogue scale) or,vertical called vertical visual analog scale usually 10 cm or 100 mm length [both the gradations are used]. It is anchored by two verbal descriptors, one for each symptom extreme.
  There could be variation in verbal descriptor anchors depending on intended use of the scale.
  For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [on 100-mm scale]
Side Effects | 4 weeks
  Gastric Pain, Constipation/Diarrhea, Blood Pressure, Dizziness, Headache, Elevated Creatinine, Bronchospasm, LFT's, Edema/Fluid Retention.
Patient Satisfaction Rate | 4 weeks
  Patient Satisfaction Rate will be determined a 5 point scale (0 -not at satisfied to 4 - completely satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Rachid Mohammad, MD, Principal Investigator — New Mazloum Hospital; Omar Tabbouche, Pharm D, Study Director — New Mazloum Hospital
Locations (1):
- New Mazloum Hospital, Tripoli, Lebanon